CLINICAL TRIAL: NCT04489446
Title: Sildenafil for Treating Patients With COVID-19 and Perfusion Mismatch: A Pilot Randomised Trial
Brief Title: Sildenafil in COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: Hospital Naval Almirante Nef, Viña del Mar, Chile (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez Lomakin, Investigator, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNAB-003
Record Dates: First submitted 2020-07-25; First posted 2020-07-28 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Covid19; SARS-COV2 Infection
Keywords: COVID19; SARS-COV2 Infection; Sildenafil; Phosphodiesterase 5 inhibitors
MeSH Terms: conditions — COVID-19 | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised to either sildenafil or placebo for up to seven days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Experimental): Patients allocated to this arm will receive Sildenafil 25mg every 8 hours orally for up to seven consecutive days.
  Interventions: Drug: Sildenafil
- Control (Placebo Comparator): Patients allocated to this arm will receive a placebo that will be similar in form to sildenafil pills in the interventional arm. These doses will be scheduled every 8 hours and wil be administered orally por up to seven consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Patients allocated to this arm will receive Sildenafil 25mg every 8 hours orally for up to seven consecutive days.
  Arms: Sildenafil
Drug: Placebo — Patients allocated to this arm will receive a matching placebo similar to Sildenafil pills used in the intervention arm. Placebos will be delivered orally every 8 hours for up to seven consecutive days.
  Arms: Control

SUMMARY:
This randomised trial aims to assess the role of sildenafil in improving oxygenation amongst hospitalised patients with COVID19.

DETAILED DESCRIPTION:
Perfusion anomalies, namely hypoperfusion of healthy lung and vasoplegia with hyperperfusion of diseased lung areas, have been recently described amongst patients with COVID19. In this triple-blind pilot randomised trial, adult patients with high clinical suspicion of SARS-CoV2 infection and perfusion defects in a substraction computed tomography angiography will be randomised in a 1:1 ratio to receive sildenafil or placebo. Informed consent will be obtained from every included participant. Patients requiring mechanical ventilation at baseline will be excluded, as will those who present a contraindication to sildenafil, previous users of sildenafil, those requiring therapy with nitrates, patients in which an order to limit therapeutic efforts has been issued, pregnant or breastfeeding women and those who decline to participate in this study. The primary outcome for this trial wil be oxygenation changes in blood gas analyses. Secondary outcomes will include clinical deterioration requiring admission to an intensive care unit, requirement of high-flow nasal cannula or invasive mechanical ventilation and overall survival. Patients will be followed-up until hospital discharge or up to fifteen days after randomisation. Statistical analyses will be undertaken by a statistician unaware of treatment allocation under the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant with high clinical suspicion of a SARS-CoV2 infection.
* Hypoperfusion of healthy lung areas in a substraction computed tomography angiography within 24 hours of admission to the hospital.

Exclusion Criteria:

* Requirement of therapy with nitrates of nitrites
* Arterial hypotension at presentation
* Recent diagnosis of coronary artery disease (<6 months)
* Acute heart failure at presentation
* Recent stroke (< 6 months)
* Chronic respiratory failure with CO2 retention
* Known hypersensitivity to sildenafil
* Advanced liver disease (Child-Pugh class B or higher)
* Users of cytochrome P450 3A4 inhibitors (Erythromycin, Ketoconazole, Itraconazole, Saquinavir)
* Pulmonary hypertension
* Chronic users of phosphodiesterase 5 inhibitors
* Requirement of invasive mechanical ventilation at baseline
* Decision to limit therapeutic efforts at baseline
* Pregnancy or lactation
* History of retinitis pigmentosa
* Known obstruction to left-ventricular outflow tract
* Unwillingness to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Arterial Oxygenation | One hour after sildenafil administration
  Mean difference in alveolar oxygen pressure to inspired oxygen fraction (Pa/Fi) ratios.
Arterial Oxygenation | Daily until the end of follow-up (up to 15 days after randomisation)
  Mean difference in alveolar oxygen pressure to inspired oxygen fraction (Pa/Fi) ratios.
Alveolo-arterial gradient | One hour after sildenafil administration
  Mean difference in the alveolo-arterial gradient between study groups.
Alveolo-arterial gradient | Daily until the end of follow-up (up to 15 days after randomisation)
  Mean difference in the alveolo-arterial gradient between study groups.

SECONDARY OUTCOMES:
Intensive care unit admission | Up to two weeks after randomisation
  Proportion of patients requiring admission to an intensive care unit in each study group
Noninvasive Mechanical Ventilation or Requirement of High-Flow Nasal Cannula | Up to two weeks after randomisation
  Proportion of patients requiring noninvasive mechanical ventilation o high-flow nasal cannula unit in each study group
Invasive mechanical ventilation | Up to two weeks after randomisation
  Proportion of patients requiring invasive mechanical ventilation in each study group
Survival | Up to two weeks after randomisation
  Proportion of patients that survived COVID19 in each study group

OTHER OUTCOMES:
Adverse events | Up to two weeks after randomisation
  Adverse events attributable to sildenafil use.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Santamarina, MD, Study Director — Hospital Naval Almirante Nef; Felipe Martinez, MD, MSc, Principal Investigator — Universidad Andres Bello
Locations (1):
- Hospital Naval Almirante Nef, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Lippi G, Plebani M. Laboratory abnormalities in patients with COVID-2019 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1131-1134. doi: 10.1515/cclm-2020-0198. No abstract available. PMID 32119647
- [Background] Santamarina MG, Boisier D, Contreras R, Baque M, Volpacchio M, Beddings I. COVID-19: a hypothesis regarding the ventilation-perfusion mismatch. Crit Care. 2020 Jul 6;24(1):395. doi: 10.1186/s13054-020-03125-9. No abstract available. PMID 32631389
- [Background] Gheblawi M, Wang K, Viveiros A, Nguyen Q, Zhong JC, Turner AJ, Raizada MK, Grant MB, Oudit GY. Angiotensin-Converting Enzyme 2: SARS-CoV-2 Receptor and Regulator of the Renin-Angiotensin System: Celebrating the 20th Anniversary of the Discovery of ACE2. Circ Res. 2020 May 8;126(10):1456-1474. doi: 10.1161/CIRCRESAHA.120.317015. Epub 2020 Apr 8. PMID 32264791
- [Background] Wu Z, Hu R, Zhang C, Ren W, Yu A, Zhou X. Elevation of plasma angiotensin II level is a potential pathogenesis for the critically ill COVID-19 patients. Crit Care. 2020 Jun 5;24(1):290. doi: 10.1186/s13054-020-03015-0. No abstract available. PMID 32503680
- [Derived] Santamarina MG, Beddings I, Lomakin FM, Boisier Riscal D, Gutierrez Claveria M, Vidal Marambio J, Retamal Baez N, Pavez Novoa C, Reyes Allende C, Ferreira Perey P, Gutierrez Torres M, Villalobos Mazza C, Vergara Sagredo C, Ahumada Bermejo S, Labarca Mellado E, Barthel Munchmeyer E, Marchant Ramos S, Volpacchio M, Vega J. Sildenafil for treating patients with COVID-19 and perfusion mismatch: a pilot randomized trial. Crit Care. 2022 Jan 3;26(1):1. doi: 10.1186/s13054-021-03885-y. PMID 34980198
- See also: COVID-19 Dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins University (JHU) — https://coronavirus.jhu.edu/map.html